CLINICAL TRIAL: NCT00004243
Title: A Phase I Study of Oxaliplatin in Combination With Docetaxel (Taxotere) Metastatic/Recurrent Solid Tumors
Brief Title: Docetaxel and Oxaliplatin in Treating Patients With Metastatic or Recurrent Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067488; U01CA062505 (NIH); CHNMC-PHASEI-24; CHNMC-IRB-99081; LAC-USC-OC-99-2; NCI-T99-0004
Record Dates: First submitted 2000-01-28; First posted 2003-04-18 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Docetaxel; Oxaliplatin

INTERVENTIONS:
Drug: docetaxel
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of docetaxel and oxaliplatin in treating patients who have metastatic or recurrent solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of docetaxel when followed by oxaliplatin in patients with metastatic or recurrent solid tumors. II. Describe the toxicities of this regimen in this patient population at each dose level studied. III. Evaluate the pharmacokinetics and pharmacodynamics of this regimen in these patients.

OUTLINE: This is a dose escalation study of docetaxel. Patients receive docetaxel IV over 1 hour followed by oxaliplatin IV over 2 hours on day 1 every 3 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Patients are followed for disease progression.

PROJECTED ACCRUAL: A total of 15-20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic or recurrent solid tumor that has failed standard therapy or for which no standard therapy exists No known brain metastases or carcinomatosis meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 OR Karnofsky 60-100% Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST/ALT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.25 times ULN Calcium no greater than 12 mg/dL Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No evidence of neuropathy No history of allergy to platinum compounds No history of allergy to antiemetics appropriate for administration in conjunction with protocol directed chemotherapy No uncontrolled concurrent illness (e.g., ongoing or active infection) No medical, social, or psychological factors that would preclude consent and follow up

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: Prior chemotherapy, including fluorouracil and cisplatin, allowed At least 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Recovered from prior surgery Other: At least 30 days since other prior investigational drugs No other concurrent investigational or commercial agents or therapies No concurrent antiretroviral therapy (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California